CLINICAL TRIAL: NCT05712785
Title: Clinical Study on the Treatment of Upper Urinary Tract Stones by Shuotong Scope
Brief Title: Shuotongo Ureteroscopy for Upper Urinary Tract Stones
Acronym: SFUUTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Handan First Hospital (Other)
Responsible Party: Principal Investigator, kunwu-yan, Research Project Leader, Handan First Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20231925-1
Record Dates: First submitted 2023-01-26; First posted 2023-02-03 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Urinary Calculi; Ureterocele
MeSH Terms: conditions — Urinary Calculi; Ureterocele

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shuotong Ureteroscopy group (Experimental): Shuotong Ureteroscopy: a ureteroscope that can lithotripsy and lithotripsy simultaneously
  Interventions: Device: Use of shuotong ureteroscopy
- Ureteroscopy group (No Intervention): Ureteroscopy group：using conventional ureteroscopy

INTERVENTIONS:
Device: Use of shuotong ureteroscopy — Treatment of patients with ureteral stones using the Shuotong-scopy
  Arms: Shuotong Ureteroscopy group

SUMMARY:
The purpose of this study is to use the Shuotong ureteroscopy for surgical treatment of patients with upper urinary tract stones, taking advantage of the fact that the Shuotong mirror can be used for simultaneous lithotripsy and stone removal, thus maximizing the discharge of stones from the body and improving the stone removal rate.

DETAILED DESCRIPTION:
Ureteroscopy via the natural lumen has the advantages of being non-invasive, safe and repeatable. This is where Shuotongo ureteroscopy, a new type of ureteroscopy, has not yet become fully popular. Usually, most patients with upper urinary tract stones are treated by ureteroscopy or with flexible ureteroscopy, because these endoscopes usually break the stones and ask the patient to drink more water to expel the stones by themselves, after the operation, it is usually easy to leave stones in the body, and some patients even form stone streets to block the ureter again after the operation. In some patients, stones may form again and obstruct the ureter again. The Shuotong Ureteroscopy has the advantages of stone crushing and stone removal, which can synchronize the process of stone crushing and stone removal and maintain a good surgical view. It has the advantages of simple operation, less trauma and high safety for the operation via natural channel, especially for the large stones in the upper urinary tract and Gantun stones.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Ureteral calculus Must be able to cooperate with the treatment

Exclusion Criteria:

* Patients had severe urinary tract infections; patients had other conditions which investigators thought not suitable for the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Stone removal rate | 1 week after surgery
  Residual stones in the body after surgery

SECONDARY OUTCOMES:
Surgery time | During surgery
  Time from start of surgery to end of surgery

CONTACTS AND LOCATIONS:
Overall Officials: kunwu yan, Master, Principal Investigator — Handan First Hospital
Locations (1):
- Kunwu Yan, Handan, Hebei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lai L, Zhang W, Zheng F, Wang T, Bai P, Liu Z, Zheng J, Shao Z, Duan B, Wang H, Xing J, Chen H, Huang Y, Chen B. Comparison of the Efficacy of ShuoTong Ureteroscopy and Simple Flexible Ureteroscopy in the Treatment of Unilateral Upper Ureteral Calculi. Front Surg. 2021 Sep 27;8:707022. doi: 10.3389/fsurg.2021.707022. eCollection 2021. PMID 34646858
- [Result] Qiao D, Cheng L, Xiaomei T, Baolei S, Yingyi L, Hui Z, Shaohua B, Wei L, U DY, Fangqiong D, Jie L, Shuangning L. Effect of ultra-mini percutaneous nephrolithotomy and ShuoTong ureteroscopy on the stress response, inflammatory indices, and urokinase level in patients with polycystic kidney disease complicated with renal calculus. Cell Mol Biol (Noisy-le-grand). 2022 Feb 4;67(5):309-316. doi: 10.14715/cmb/2021.67.5.42. PMID 35818238
- [Result] Gan S, Guo Z, Zou Q, Gu C, Xiang S, Li S, Ye Z, Wang S. Diagnosis accuracy of PCA3 level in patients with prostate cancer: a systematic review with meta-analysis. Int Braz J Urol. 2020 Sep-Oct;46(5):786-793. doi: 10.1590/S1677-5538.IBJU.2019.0521. PMID 32539255